CLINICAL TRIAL: NCT00995761
Title: Phase II Study of Biweekly Schedule of Docetaxel and Cisplatin in High Risk Patients With Unresectable Non-small Cell Lung Cancer
Brief Title: Biweekly Schedule of Docetaxel and Cisplatin in High Risk Patients With Unresectable Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gyeongsang National University Hospital (Other)
Responsible Party: Principal Investigator, Gyeong-Won Lee, Associate professor, Gyeongsang National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GNUHIRB-2009-30
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Results first posted 2014-03-03 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: biweekly; docetaxel; cisplatin; non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- biweekly schedule (No Intervention): docetaxel 40mg/m2 on day 1,15 every 4weeks cisplatin 40mg/m2 on day 1,15 every 4weeks
  Interventions: Drug: Docetaxel and Cisplatin

INTERVENTIONS:
Drug: Docetaxel and Cisplatin — splitted administration of docetaxel and cisplatin.
  Other Names: Docetaxel (Sanofi-Aventis); Cisplatin

SUMMARY:
The rationale of phase II study of biweekly docetaxel and cisplatin in patients with unresectable NSCLC are follows:

First, the optimal dose and schedule of combination with docetaxel and cisplatin are still controversial (3 weekly versus weekly).

Platinum-based combination chemotherapy improves the survival of patients with advanced non-small cell lung cancer (NSCLC) in the first-line setting.

Combination chemotherapy with docetaxel and cisplatin is one of the standard platinum-based regimens for treating NSCLC. However, usual standard 3 weekly regimen with docetaxel and cisplatin have consistently produced frequent Grade 3-4 neutropenia, and febrile neutropenia.

Although weekly docetaxel and cisplatin is better tolerated than chemotherapy every 3 weeks, especially in the first line setting in terms of myelosuppression, the optimal dose and schedule for administration of the two drugs has not yet been determined.

Both 3-weekly docetaxel plus cisplatin and weekly schedule showed similar response rates but had different toxicity profiles. The most frequent grade 3 or 4 toxicities were neutropenia in the 3 weekly schedule and fatigue or asthenia in the weekly schedule.

Second, docetaxel and cisplatin have different action and mechanism. Docetaxel showed characteristic early bone marrow suppression 5-7 days after infusion compared with usual 14 days after infusion of cisplatin. Thus, nadir period is not overlapped when the investigators administered both drugs concomittantly.

Third, there are many feasible reports of biweekly administration of docetaxel in patients with NSCLC, breast cancer, stomach cancer, and ovarian cancer with better safety profiles.

Therefore,the investigators designed this phase II study to evaluate the efficacy and toxicity of biweekly schedule of docetaxel and cisplatin in patients with unresectable NSCLC and test the hypothesis that biweekly schedule of docetaxel and cisplatin is better tolerated than both standard 3 week and weekly schedule in terms of hematologic (neutropenia) and non-hematologic toxicities (asthenia, interstitial pneumonitis. Additionally the investigators will evaluate polymorphism associated with this study.

DETAILED DESCRIPTION:
Study design is followings: The sample size was calculated according to Simon's two stage optimal design. Assuming a response rate of 40%, a probability of error of 5% and a power of 80%, a total of 48 patients (43 patients plus 5 patients to compensate a 10% drop-out rate) were enrolled. In the initial stage, 13 evaluable patients were to be entered into the study and evaluated for their response. If ≥ 3 responses were observed during the first stage, then 30 additional patients were to be entered in the second stage. The statistical evaluation was performed based on the intention to-treat analysis.

The combination chemotherapy consisted of docetaxel of 40mg/m2 as a 1-hour infusion followed by cisplatin 40mg/m2 as a 30-minutes intravenous infusion and both drugs were given on days 1, and 15 in an outpatient setting. Patients also received adequate hydration with at least 1,500ml of half saline or normal saline before cisplatin administration. All the patients received antiemetic therapy that consisted of intravenous 5-HT3 antagonist and dexamethasone before docetaxel administration. The treatment cycles were repeated every 4 weeks until the maximum six cycles.

The patients whose absolute neutrophil count and platelet count were greater than or equal to 1.500 and 100,000/mm3, respectively, and who had lower than or equal to grade 1 non-hematologic toxicity (excluding alopecia) received chemotherapy on day 1 of each cycle.

On days 15 of each cycle, the minimum requirements to receive chemotherapy were an absolute neutrophil count between 1000 and 1,500/mm3, a platelet count ≥75,000/mm3 and no grade ≥2 nonhematologic toxicity (excluding alopecia).

If these conditions were not met on days 1, or 15, then chemotherapy was postponed for 1 week. A delay of more than 3 weeks resulted in withdrawal from the study.

If there were any grade 3 to 4 hematologic toxicities at the nadir of the previous cycle, or febrile neutropenia with or without documented infection, then administration of both drugs in the subsequent cycles was reduced by 25% from the planned dose.

The Administration of granulocyte-colony stimulating factor (G-CSF) was allowed in the presence of febrile neutropenia, and grade 3 or 4 neutropenia.

In the presence of grade 3 or 4 non-hematologic toxicity (except nausea, vomiting and alopecia), the treatment was postponed until resolution of the toxicity and then both drug doses were reduced by 25% for the next cycle. Treatment was stopped at any time for documented disease progression, unacceptable toxicity or according to the patient's own refusal.

The pretreatment baseline evaluation included a complete medical history and physical examination, a complete blood cell count (CBC) with the differentials, chemistry profiles and performance status. Chest X-rays, chest and upper abdominal computed tomography (CT) scans, brain CT scan or magnetic resonance imaging, a radionuclide bone scan and other diagnostic procedures were performed as clinically indicated.

During treatment, a limited history taking, physical examination, assessment of toxicity, a complete blood cell count with the differentials and blood chemistry tests were repeated weekly. A chest X-ray was performed every 4 weeks before each cycle.

Appropriate imaging studies, including CT scans of the chest and upper abdomen, were performed every two cycles to assess the treatment response, and sooner if needed for documenting disease progression. The objective tumor responses were assessed according to the RECIST criteria. The response rate was calculated as the ratio of the number of patients who achieved a complete or partial response to the number of enrolled patients. Overall survival (OS) and Time to progression (TTP) were calculated from the start of therapy until death and progression, respectively, or until the last follow-up. Toxicities were evaluated according to the National Cancer Institute Common Toxicity Criteria (NCI-CTC) scale version 3.0.

ELIGIBILITY:
Inclusion Criteria:

* patients who were≥ 65 years of age and they had an Easten Cooperative Oncology Group (ECOG) performance status (PS) of 0-2, or the patients who were < 65 years of age and they had an ECOG PS 2
* histologically confirmed non-small cell carcinoma
* stages IIIB-IV disease
* adequate hematologic parameters (hemoglobin concentration of at least 9.0 g/dL, absolute neutrophil count ≥1,500/mm3, and platelet count ≥100,000/mm3), renal function (serum creatinine ≤1.5 mg/dL), and liver function (total bilirubin ≤1.5 mg/dL and serum transaminase level less than twice the upper limit of normal)
* at least one bi-dimensionally measurable lesion, according to the Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1

Exclusion Criteria:

* Active infection
* Prior chemotherapy, radiotherapy or surgery for their disease,
* A history of myocardial infarction in the last 3 months before entry to the study
* Uncontrolled congestive heart failure or hypertension
* Uncontrolled diabetes mellitus, pregnancy, lactation or a prior second primary cancer except for cervix cancer in situ or skin cancer
* All the patients provided written informed consent before they entered the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gyeong-Won Lee, M.D.Ph.D., Principal Investigator — Gyeongsang National University Hospital IRB
Locations (1):
- Gyeongsang National University Hospital, Jinju, Gyeongsang-Nam-Do, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: anticipated dates of final recruitment: September 2011 Type of location: University Hospital Clinic
Pre-assignment Details: not specific problems
Period: Overall Study
Arm/Group | Biweekly Schedule
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Biweekly Schedule
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 25
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 66 (1.5) [61 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 43
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 48

OUTCOME MEASURES:

1. Primary Outcome: Response Rates Confirmed With CT or MRI
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
  During treatment, a limited history, physical examination, assessment of toxicity, CBC with differentials, and blood chemistry tests were repeated weekly. A chest X-ray was performed every 2 weeks before each cycle. Appropriate imaging studies, including CT scans of the chest and upper abdomen, were performed every two cycles to assess the treatment response, and sooner, if required, to document disease progression. Objective tumor responses were assessed according to the RECIST criteria V 1.0.
Time Frame: after every 2 cycles of docetaxel and cisplatin
Population: The sample size was calculated according to Simon's two-stage optimal design.The statistical evaluation was performed based on an ITT analysis. Descriptive statistics are reported as proportions and medians. OS and TTP were assessed by the K-M method, and the 95% CI for the median time to events was computed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Biweekly Schedule of Docetaxel and Cisplatin: we conducted the present phase II study to investigate the efficacy and safety of a biweekly schedule of docetaxel and cisplatin in patients with unresectable NSCLC.
Arm/Group | Biweekly Schedule of Docetaxel and Cisplatin
Number analyzed (Participants) | 48
percentage of participants | 64.6 [52.1 to 77.1]

2. Secondary Outcome: Time to Progression and Overall Survival Confirmed Through Follow-up and Observation Following Treatment
Time Frame: From date of enrollment in this study until the date of first documented progression or date of death from any cause, whichever came first, after every 2 cycles of docetaxel and cisplatin
Reporting Status: Not Posted

3. Primary Outcome: We Conducted the Present Phase II Study to Investigate the Efficacy and Safety of a Biweekly Schedule of Docetaxel and Cisplatin in Patients With Unresectable NSCLC.
Description: we conducted the present phase II study to investigate the efficacy and safety of a biweekly schedule of docetaxel and cisplatin in patients with unresectable NSCLC (OS, TTP, and Others)
Time Frame: after every 2 cycles of docetaxel and cisplatin
Reporting Status: Not Posted, anticipated posting 2012-12
Measure: Median

ADVERSE EVENTS:
Arm/Group | Biweekly Schedule
Serious Adverse Events (participants affected / at risk) | 7/48
Other Adverse Events (participants affected / at risk) | 0/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biweekly Schedule (N=48)
Diarrhea (Gastrointestinal disorders) | 5 (5) — Diarrhea, Grade 3 : 4 patients(8.3)
neutropenia (Blood and lymphatic system disorders) | 3 (3) — Anemia, Grade 3: 7 patients (14.5)
leukopenia (Blood and lymphatic system disorders) | 4 (4) — Leukopenia, grade 3: 4 patients (8.3)
Infection (Infections and infestations) | 5 (5) — Infection, Grade 3: 5 patients (10.4)
Asthenia (Musculoskeletal and connective tissue disorders) | 3 (3) — Asthenia, Grade 3: 3 patients (6.3)
anemia (Blood and lymphatic system disorders) | 7 (7) — Anemia, Grade 3: 7 patients (14.5)

LIMITATIONS AND CAVEATS:
completed without a major limitation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No